CLINICAL TRIAL: NCT00087646
Title: A Randomized, Open-label Study of the Effect of PEGASYS Combined With Ribavirin on Sustained Virologic Response in Patients With Chronic Hepatitis C Who Did Not Respond to Previous Pegintron/Ribavirin Combination Therapy
Brief Title: REPEAT Study - A Study of PEGASYS (Peginterferon Alfa-2a (40KD)) Therapy in Combination With COPEGUS (Ribavirin) in Patients With Chronic Hepatitis C (CHC) Who Did Not Respond to Previous PegIntron (Peginterferon Alfa-2b (12KD))/Ribavirin Combination Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MV17150
Record Dates: First submitted 2004-07-12; First posted 2004-07-14 (Estimated); Results first posted 2016-01-14 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2015-12

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; peginterferon alfa-2a

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: Ribavirin; Drug: peginterferon alfa-2a [Pegasys]
- 2 (Experimental)
  Interventions: Drug: Ribavirin; Drug: peginterferon alfa-2a [Pegasys]
- 3 (Experimental)
  Interventions: Drug: Ribavirin; Drug: peginterferon alfa-2a [Pegasys]
- 4 (Active Comparator)
  Interventions: Drug: Ribavirin; Drug: peginterferon alfa-2a [Pegasys]

INTERVENTIONS:
Drug: Ribavirin — 1000/1200mg po daily for 72 weeks
  Arms: 1; 3
Drug: Ribavirin — 1000/1200mg po daily for 48 weeks
  Arms: 2; 4
Drug: peginterferon alfa-2a [Pegasys] — 360 micrograms sc weekly for 12 weeks, followed by 180 micrograms sc weekly for 60 weeks
  Arms: 1
Drug: peginterferon alfa-2a [Pegasys] — 360 micrograms sc weekly for 12 weeks, followed by 180 micrograms sc weekly for 36 weeks.
  Arms: 2
Drug: peginterferon alfa-2a [Pegasys] — 180 micrograms sc weekly for 72 weeks
  Arms: 3
Drug: peginterferon alfa-2a [Pegasys] — 180 micrograms sc weekly for 48 weeks
  Arms: 4

SUMMARY:
This 4 arm study is designed for patients with CHC who have not responded to peginterferon alfa-2b (12KD)/ribavirin combination therapy. In these patients, the effects of lengthening the duration of treatment, as well as including an initial 12-week period of high-dose PEGASYS (360 micrograms sc), are compared with the standard combination therapy of PEGASYS (180 micrograms sc) and ribavirin (1000-1200mg po). The anticipated time on study treatment is 1-2 years and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >=18 years of age;
* CHC infection;
* liver biopsy (in <24 calendar months of first dose), with results consistent with CHC infection;
* use of 2 forms of contraception during study and 6 months after the study in both men and women;
* Lack of response to previous treatment with peginterferon alfa-2b (12KD)/ribavirin combination therapy given for >=12 weeks.

Exclusion Criteria:

* women who are pregnant or breastfeeding;
* male partners of women who are pregnant;
* conditions associated with decompensated liver disease;
* other forms of liver disease, including liver cancer;
* human immunodeficiency virus infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 948 (Actual)
Dates: Start 2003-09; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (94):
- United States (33):
  - Mobile, Alabama
  - Scottsdale, Arizona
  - Los Angeles, California
  - Pasadena, California
  - San Diego, California
  - Ukiah, California
  - Farmington, Connecticut
  - Bradenton, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Atlanta, Georgia
  - Savannah, Georgia
  - Chicago, Illinois
  - Des Moines, Iowa
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Minneapolis, Minnesota
  - Rochester, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - Florham Park, New Jersey
  - Albuquerque, New Mexico
  - Williamsville, New York
  - Lancaster, Pennsylvania
  - Philadelphia, Pennsylvania
  - Cranston, Rhode Island
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Burlington, Vermont
  - Richmond, Virginia
- Belgium (3):
  - Brussels
  - Ghent
  - Leuven
- Rio de Janeiro, Brazil
- Canada (2):
  - Vancouver, British Columbia
  - Toronto, Ontario
- France (9):
  - Clichy
  - Créteil
  - Lille
  - Lyon
  - Marseille
  - Montpellier
  - Paris
  - Pessac
  - Toulouse
- Germany (18):
  - Berlin
  - Bochum
  - Bonn
  - Cologne
  - Düsseldorf
  - Erlangen
  - Frankfurt am Main
  - Freiburg im Breisgau
  - Hamburg
  - Hanover
  - Heidelberg
  - Homburg/saar
  - Kassel
  - Kiel
  - Mainz
  - München
  - Oberhausen
  - Würzburg
- Greece (3):
  - Alexandroupoli
  - Athens
  - Thessaloniki
- Italy (7):
  - Bari
  - Bologna
  - Milan
  - Padua
  - Palermo
  - Roma
  - Torino
- Portugal (2):
  - Coimbra
  - Lisbon
- Spain (8):
  - Alicante
  - Barcelona
  - Granada
  - Madrid
  - Málaga
  - Santander
  - Seville
  - Valencia
- Sweden (3):
  - Gothenburg
  - Huddinge
  - Lund
- Zurich, Switzerland
- Turkey (Türkiye) (3):
  - Ankara
  - Istanbul
  - Izmir
- Birmingham, United Kingdom

REFERENCES:
- [Derived] Marcellin P, Craxi A, Brandao-Mello CE, Di Bisceglie AM, Andreone P, Freilich B, Rajender Reddy K, Olveira Martin A, Teuber G, Messinger D, Hooper G, Wat C, Tatsch F, Jensen DM. Predicting early and sustained virological responses in prior nonresponders to pegylated interferon alpha-2b plus ribavirin retreated with peginterferon alpha-2a plus ribavirin and the benefit-risk ratio of retreatment. J Clin Gastroenterol. 2013 Oct;47(9):786-93. doi: 10.1097/MCG.0b013e31827b9b45. PMID 23442834
- See also: This is a full publication titled Re-treatment of Patients With Chronic Hepatitis C Who Do Not Respond to Peginterferon- alfa2b, A Randomized Trial — http://www.ncbi.nlm.nih.gov/pubmed/19380853

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 16 September 2003 to 27 February 2007. Participants were recruited over a total of 106 centers [(United States (37), Germany (19), Spain (10), France (9), Italy (7), Greece (5), Turkey (4), Belgium (3), Canada (3), Portugal (3), Sweden (3), Brazil (1), Switzerland (1), and UK (1)] in the study.
Pre-assignment Details: A total of 950 participants were randomized (318, 158, 158, and 316 in groups A, B, C, and D, respectively), 942 received the study medication. A total of 8 randomized participants did not receive study drug for various reasons which includes withdrew consent (5), violated the study entry criteria (1), and two had other protocol violations.
Groups:
- Group A: Participants received 360 microgram (mcg) of peginterferon alfa-2a (PEG-IFN alfa-2a) once weekly plus 1000/1200 mg of ribavirin daily for 12 weeks, and thereafter 180 mcg of PEG-IFN alfa-2a once weekly plus 1000/1200 mg of ribavirin daily for 60 weeks.
- Group B: Participants received 360 mcg of PEG-IFN alfa-2a once weekly plus 1000/1200 mg of ribavirin daily for 12 weeks, and thereafter 180 mcg of PEG-IFN alfa-2a once weekly plus 1000/1200 mg of ribavirin daily for 36 weeks.
- Group C: Participants received 180 mcg of PEG-IFN alfa-2a once weekly plus 1000/1200 mg of ribavirin daily for 72 weeks.
- Group D: Participants received 180 mcg of PEG-IFN alfa-2a once weekly plus 1000/1200 mg of ribavirin daily for 48 weeks.
Period: Overall Study
Arm/Group | Group A | Group B | Group C | Group D
Started | 317 | 156 | 156 | 313
Completed | 182 | 114 | 91 | 229
Not Completed | 135 | 42 | 65 | 84
Not completed — Adverse Event | 37 | 6 | 18 | 20
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 1 | 2 | 2
Not completed — Insufficient therapeutic response | 64 | 24 | 38 | 51
Not completed — Refused Treatment/Did Not Cooperate | 13 | 6 | 4 | 5
Not completed — Failure to Return | 5 | 2 | 2 | 3
Not completed — Administrative/Other | 6 | 1 | 1 | 2
Not completed — Other Protocol Violation | 3 | 1 | 0 | 0
Not completed — Violation of Selection Criteria at Entry | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat analysis population (ITT) included, all participants randomized who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Group D | Total
Number analyzed (Participants) | 317 | 156 | 156 | 313 | 942
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (8.73) | 48.8 (9.93) | 49.4 (8.46) | 48.5 (8.97) | 48.6 (8.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 62 | 49 | 101 | 326
  Male | 203 | 94 | 107 | 212 | 616

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sustained Virological Response Rate
Description: Sustained Virological Response (SVR) was defined as the percentage of participants with a undetectable hepatitis C virus- ribonucleic acid (HCV RNA) 24 weeks after the end of the treatment period (defined as a single last HCV RNA < 50 International Units Per Millilitre (IU/mL) measured >= 20 weeks after treatment end, ie, >=140 days after treatment end.
Time Frame: Up to 72 weeks (Group A) and 48 weeks (Group D)
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Group A | Group D
Number analyzed (Participants) | 317 | 313
participants | 52 | 27
Statistical Analysis 1: Comparison: Group A vs Group D; Group A Vs Group D; Test type: Superiority or Other; p = 0.0060, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.00, 95% CI 2-sided [1.21 to 3.31]

2. Secondary Outcome: Number of Participants With Sustained Virological Response (Groups A + B vs Groups C + D)
Description: SVR was defined as the percentage of participants with a undetectable hepatitis C virus- ribonucleic acid (HCV RNA) 24 weeks after the end of the treatment period (defined as a single last HCV RNA < 50 International Units Per Millilitre (IU/mL) measured >= 20 weeks after treatment end, ie, >=140 days after treatment end.
Time Frame: At Week 48 and Week 72
Population: ITT population included all participants randomized who received at least one dose of study medication.
Measure: Number; unit: participants
Groups:
- Group A + Group B: Group A - Participants received 360 microgram (mcg) of peginterferon alfa-2a (PEG-IFN alfa-2a) once weekly plus 1000/1200 mg of ribavirin daily for 12 weeks, and thereafter 180 mcg of PEG-IFN alfa-2a once weekly plus 1000/1200 mg of ribavirin daily for 60 weeks.
  Group B - Participants received 360 mcg of PEG-IFN alfa-2a once weekly plus 1000/1200 mg of ribavirin daily for 12 weeks, and thereafter 180 mcg of PEG-IFN alfa-2a once weekly plus 1000/1200 mg of ribavirin daily for 36 weeks.
- Group C + Group D: Group C - Participants received 180 mcg of PEG-IFN alfa-2a once weekly plus 1000/1200 mg of ribavirin daily for 72 weeks.
  Group D - Participants received 180 mcg of PEG-IFN alfa-2a once weekly plus 1000/1200 mg of ribavirin daily for 48 weeks.
Arm/Group | Group A + Group B | Group C + Group D
Number analyzed (Participants) | 473 | 469
participants | 63 | 49
Statistical Analysis 1: Comparison: Group A + Group B vs Group C + Group D; Test type: Superiority or Other; p = 0.9228, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.63 to 1.51]

3. Secondary Outcome: Number of Participants With Sustained Virological Response (Groups A + C vs Groups B + D)
Description: as for outcome 2
Time Frame: At Week 48 and Week 72
Population: ITT population included all participants randomized who received at least one dose of study medication.
Measure: Number; unit: participants
Groups:
- Group A + Group C: Group A - Participants received 360 microgram (mcg) of peginterferon alfa-2a (PEG-IFN alfa-2a) once weekly plus 1000/1200 mg of ribavirin daily for 12 weeks, and thereafter 180 mcg of PEG-IFN alfa-2a once weekly plus 1000/1200 mg of ribavirin daily for 60 weeks.
  Group C - Participants received 180 mcg of PEG-IFN alfa-2a once weekly plus 1000/1200 mg of ribavirin daily for 72 weeks.
- Group B + Group D: Group B - Participants received 360 mcg of PEG-IFN alfa-2a once weekly plus 1000/1200 mg of ribavirin daily for 12 weeks, and thereafter 180 mcg of PEG-IFN alfa-2a once weekly plus 1000/1200 mg of ribavirin daily for 36 weeks.
  Group D - Participants received 180 mcg of PEG-IFN alfa-2a once weekly plus 1000/1200 mg of ribavirin daily for 48 weeks.
Arm/Group | Group A + Group C | Group B + Group D
Number analyzed (Participants) | 473 | 469
participants | 74 | 38
Statistical Analysis 1: Comparison: Group A + Group C vs Group B + Group D; Test type: Superiority or Other; p = 0.0006, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.22, 95% CI 2-sided [1.40 to 3.52]

4. Secondary Outcome: Percentage of Participants With Undetectable HCV-RNA
Description: The percentage of participants with a undetectable HCV RNA 24 weeks after the end of the treatment period (defined as a single last HCV RNA < 50 IU/mL measured >= 20 weeks after treatment end, ie, >=140 days after treatment end) are reported.
  End-of-treatment (EOT) virological response is defined as last HCV RNA measurement that is not detectable (<50 IU/mL) at study day of last dose of study medication (+/- 28 days).
Time Frame: At Week 12, 24, 48 and EOT
Population: ITT population included all participants randomized who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Group A | Group D
Number analyzed (Participants) | 317 | 313
percentage of participants
  At Week 12 | 24 | 11
  At Week 24 | 32 | 27
  At Week 48 | 32 | 26
  At EOT | 31 | 28
Statistical Analysis 1: Comparison: Group A vs Group D; At Week 12; Test type: Superiority or Other; p < .0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.64, 95% CI 2-sided [1.66 to 4.18]
Statistical Analysis 2: Comparison: Group A vs Group D; At Week 24; Test type: Superiority or Other; p = 0.1955, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.89 to 1.79]
Statistical Analysis 3: Comparison: Group A vs Group D; At Week 48; Test type: Superiority or Other; p = 0.0883, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.95 to 1.93]

5. Secondary Outcome: Percentage of Participants With >=2log Drop in HCV-RNA
Description: Reduction in HCV-RNA titers of at least 2 log10 after 12/24 weeks of study treatment (i.e. 99% reduction of viral load) was analyzed. Percentage of participants with at least a 2 log10 drop of HCV-RNA at study week 12 and 24 (lower limit of quantitation 600 IU/mL) as compared to baseline or non-detectable HCV-RNA (lower limit of detection 50 IU/mL) were reported.
Time Frame: At Week 12 and 24
Population: ITT population included all the participants randomized who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Group A | Group D
Number analyzed (Participants) | 317 | 313
percentage of participants
  Week 12 | 62 | 42
  Week 24 | 51 | 47
Statistical Analysis 1: Comparison: Group A vs Group D; Groups A vs Groups D (Week 12); Test type: Superiority or Other; p < .0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.31, 95% CI 2-sided [1.67 to 3.19]
Statistical Analysis 2: Comparison: Group A vs Group D; Groups A vs Groups D (Week 24); Test type: Superiority or Other; p = 0.3389, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.85 to 1.60]

6. Secondary Outcome: Change From Baseline in Reduction of HCV Viremia (Groups A + B vs Groups C + D)
Description: The mean change from baseline in HCV RNA level (reduction in viral load) at Week 12 and 24 were determined. HCV RNA result were not detectable (<50 IU/ML) and not quantifiable (<600 IU/ML). Baseline value were assessed on Day 1 before the administration of the first dose of study drug.
Time Frame: At Week 12 and 24
Population: ITT population included all participants randomized who received at least one dose of study medication.
Measure: Mean (95% Confidence Interval); unit: IU/ML
Arm/Group | Group A + Group B | Group C + Group D
Number analyzed (Participants) | 473 | 469
IU/ML
  HCV RNA Change from BL to Week 12 (n= 424, 421) | -2.75 [-2.89 to -2.61] | -2.18 [-2.32 to -2.03]
  HCV RNA Change from BL to Week 24 (n= 390, 399) | -2.88 [-3.05 to -2.70] | -2.64 [-2.81 to -2.47]

7. Secondary Outcome: Percentage of Participants With Maintenance of Actual End-of-Treatment Virological Response
Description: Maintenance of end-of-treatment virological response was assessed based on all participants treated and according to the actual treatment period (backward imputation method). The percentage of participants who maintained their end-of-treatment virological response was determined. Maintenance of actual end-of-treatment virological response was calculated by dividing the number of participants with a virological response both at the end of the actual untreated follow-up period and at the end of the actual treatment period by the number of participants with a virological response at the actual end of treatment.
Time Frame: Week 96 (Group A and C) and Week 72 (Group B and D)
Population: ITT population included all participants randomized who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 317 | 156 | 156 | 313
percentage of participants | 51 | 22 | 41 | 33

8. Secondary Outcome: Percentage of Participants With Relapse After End of Treatment
Description: The percentage of participants who relapsed (loss of response) after having achieved a virological response at the end of treatment was determined.
Time Frame: Week 96 (Group A and C) and Week 72 (Group B and D)
Population: ITT population included all participants randomized who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 317 | 156 | 156 | 313
percentage of participants | 49 | 78 | 59 | 67

ADVERSE EVENTS:
Time Frame: Up to Week 96 (Groups A and C) and 72-week (Groups B and D)
Description: Serious adverse events and non-serious adverse events are reported in Safety Analysis Set, which consists of all participants who received at least one dose of study medication and had a safety assessment performed post baseline.
Arm/Group | Group A | Group B | Group C | Group D
Serious Adverse Events (participants affected / at risk) | 33/317 | 14/156 | 28/156 | 33/313
Other Adverse Events (participants affected / at risk) | 306/317 | 151/156 | 150/156 | 298/313
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=317) | Group B (N=156) | Group C (N=156) | Group D (N=313)
Pneumonia (Infections and infestations) | 4 | 1 | 2 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 4
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1
Enterococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Infected insect bite (Infections and infestations) | 0 | 1 | 0 | 0
Infective spondylitis (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Osteomyelitis chronic (Infections and infestations) | 0 | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 2 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Oesophageal varices Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mallory-weiss syndrome (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lymphatic system neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Renal cell carcinoma stage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Unspecified Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 2 | 2 | 0 | 0
Aggression (Psychiatric disorders) | 1 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 1
Depression suicidal (Psychiatric disorders) | 0 | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 1
Diabetic retinopathy (Eye disorders) | 0 | 0 | 0 | 1
Retinal artery embolism (Eye disorders) | 0 | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 1 | 0
Retinal exudates (Eye disorders) | 1 | 0 | 0 | 0
Retinal vein occlusion (Eye disorders) | 0 | 0 | 1 | 0
Ulcerative keratitis (Eye disorders) | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Insulin-dependent Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 2 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 0 — General disorders and Administration site conditions
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0
Facial palsy (Nervous system disorders) | 1 | 0 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 0 | 0 | 0
Ruptured cerebral aneurysm (Nervous system disorders) | 0 | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Varicocele (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Raynaud's phenomenon (Vascular disorders) | 0 | 0 | 1 | 0
Spondylolisthesis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Sarcoidosis (Immune system disorders) | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=317) | Group B (N=156) | Group C (N=156) | Group D (N=313)
Fatigue (General disorders) | 134 | 62 | 57 | 137
Asthenia (General disorders) | 88 | 43 | 49 | 89
Pyrexia (General disorders) | 81 | 44 | 33 | 74
Influenza like illness (General disorders) | 87 | 39 | 37 | 80
Irritability (General disorders) | 54 | 32 | 27 | 54
Chills (General disorders) | 47 | 29 | 19 | 38
Pain (General disorders) | 22 | 10 | 12 | 20
Injection site erythema (General disorders) | 21 | 10 | 8 | 14
Nausea (Gastrointestinal disorders) | 91 | 50 | 41 | 78
Diarrhoea (Gastrointestinal disorders) | 66 | 31 | 27 | 44
Vomiting (Gastrointestinal disorders) | 34 | 14 | 13 | 28
Abdominal pain upper (Gastrointestinal disorders) | 30 | 11 | 10 | 32
Dyspepsia (Gastrointestinal disorders) | 16 | 9 | 10 | 19
Abdominal pain (Gastrointestinal disorders) | 18 | 8 | 11 | 15
Dry mouth (Gastrointestinal disorders) | 20 | 15 | 6 | 12
Constipation (Gastrointestinal disorders) | 12 | 6 | 6 | 17
Myalgia (Musculoskeletal and connective tissue disorders) | 70 | 46 | 39 | 80
Arthralgia (Musculoskeletal and connective tissue disorders) | 76 | 29 | 31 | 57
Back pain (Musculoskeletal and connective tissue disorders) | 31 | 18 | 8 | 39
Muscle spasms (Musculoskeletal and connective tissue disorders) | 24 | 5 | 8 | 20
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 15 | 8 | 9 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 7 | 4 | 16
Pruritus (Skin and subcutaneous tissue disorders) | 85 | 38 | 39 | 83
Alopecia (Skin and subcutaneous tissue disorders) | 53 | 31 | 27 | 43
Dry skin (Skin and subcutaneous tissue disorders) | 38 | 24 | 27 | 38
Rash (Skin and subcutaneous tissue disorders) | 37 | 24 | 14 | 43
Headache (Nervous system disorders) | 117 | 68 | 56 | 123
Dizziness (Nervous system disorders) | 32 | 15 | 17 | 29
Disturbance in attention (Nervous system disorders) | 14 | 10 | 8 | 17
Tremor (Nervous system disorders) | 9 | 8 | 3 | 8
Insomnia (Psychiatric disorders) | 99 | 46 | 47 | 89
Depression (Psychiatric disorders) | 56 | 20 | 29 | 58
Anxiety (Psychiatric disorders) | 21 | 5 | 12 | 23
Sleep disorder (Psychiatric disorders) | 14 | 9 | 7 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 62 | 26 | 33 | 64
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 33 | 19 | 19 | 44
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 24 | 9 | 6 | 15
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 | 5 | 8 | 10
Anaemia (Blood and lymphatic system disorders) | 48 | 32 | 27 | 31
Neutropenia (Blood and lymphatic system disorders) | 33 | 17 | 13 | 22
Thrombocytopenia (Blood and lymphatic system disorders) | 20 | 11 | 6 | 8
Decreased appetite (Metabolism and nutrition disorders) | 70 | 25 | 28 | 61
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 18 | 5 | 2 | 16
Sinusitis (Infections and infestations) | 17 | 6 | 5 | 12
Bronchitis (Infections and infestations) | 17 | 8 | 7 | 8
Upper respiratory tract Infection (Infections and infestations) | 15 | 8 | 11 | 5
Nasopharyngitis (Infections and infestations) | 12 | 11 | 3 | 11
Weight decreased (Investigations) | 31 | 6 | 15 | 17
Hypertension (Vascular disorders) | 21 | 11 | 8 | 12
Vision blurred (Eye disorders) | 15 | 8 | 6 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.